CLINICAL TRIAL: NCT00939874
Title: Switch From Tenofovir to Raltegravir for Low Bone Mineral Density
Acronym: TROP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St Vincent's Hospital, Sydney (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Holdsworth House Medical Practice (Other); The Alfred (Other)
Responsible Party: Principal Investigator, Andrew Carr, Professor, Head Clinical Research program, St Vincent's Hospital, Sydney
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TROP
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Results first posted 2015-06-12 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-05

CONDITIONS: HIV; Osteopenia; Osteoporosis; HIV Infections
Keywords: HIV+; Raltegravir; Tenofovir; osteopenia; osteoporosis; bone markers; treatment experienced
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis; HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Raltegravir (Experimental)
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — Raltegravir tablet 400mg is taken orally, twice daily with or without food for 48 weeks.
  Other Names: Isentress; MK-0518

SUMMARY:
The purpose of this study is to determine if low bone mineral density (a measurement of how thick and strong bones are) improves in adults with HIV infection who switch their HIV medication tenofovir to another HIV medication raltegravir.

Hypothesis:That Bone Mineral Density (BMD) will improve in osteopenic or osteoporotic patients switching from ART including tenofovir disoproxil fumarate (TDF) and a ritonavir-boosted protease inhibitor (r/PI) to ART including RAL+r/PI.

ELIGIBILITY:
Inclusion Criteria:

1. provision of written, informed consent
2. HIV-infected adults at least 18 years of age
3. receiving stable ART including TDF and a r/PI for the previous 6 months
4. no prior PI genotypic resistance or known replication of HIV in patients receiving a PI
5. plasma HIV RNA < 50 copies/ml for at least the previous 3 months
6. spine or neck of femur t-score ≤ -1.0 (i.e. WHO-defined osteopenia) measured by dual energy x-ray absorptiometry (DEXA)

   Exclusion Criteria:
7. participation in any other clinical trial (unless approved by the study PI)
8. use of TDF for previously active chronic hepatitis B infection
9. receiving or requiring therapy for low BMD (including prior fragility fracture)
10. using oral corticosteroids or inhaled fluticasone
11. virological failure on, or intolerance to, RAL
12. contra-indication to RAL therapy (see appendix 2)
13. breast-feeding
14. pregnancy
15. secondary, endocrinological cause of low BMD:25-hydroxy vitamin D deficiency, hypogonadism: a)symptomatic b)asymptomatic defined by total testosterone > 25% below lower limit of reference range and/or luteinizing hormone > 2 x upper limit of normal (ULN),untreated hypothyroidism or hyperparathyroidism according to local reference ranges

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-10; Primary Completion 2012-06 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Carr, Professor, Principal Investigator — St Vincents Hospital
Locations (4):
- Australia (4):
  - East Sydney Doctors, Sydney, New South Wales
  - Holdsworth Medical Practice, Sydney, New South Wales
  - St Vincents Hospital, Sydney, New South Wales
  - The Alfred Hospital, Melbourne, Victoria

RESULTS

PARTICIPANT FLOW:
Groups:
- Raltegravir: Thirty seven adults receiving tenofovir (TDF) and a ritonavir-boosted protease inhibitor (r/PI) were switched from TDF to raltegravir (RAL) in this open-label, non-randomised trial. Raltegravir tablet 400mg was taken orally, twice daily for 48 weeks
Period: Overall Study
Arm/Group | Raltegravir
Started | 52
Completed Week 48 | 37
Completed | 32
Not Completed | 20

BASELINE CHARACTERISTICS:
Arm/Group | Raltegravir
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 50 [30 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 36
Region of Enrollment [Number; unit: participants]
  Australia | 37

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Bone Mineral Density (BMD) of Lumbar Spine and Hips
Description: Percent Change in Bone Mineral Density of Lumbar Spine and Hips from Baseline to Weeks 48 and 96
Time Frame: from Baseline to Weeks 48 and 96
Population: Week 48 data were available for 37 completed participants and Week 96 data were available for 32 completed participants. Fifteen of the enrolled 52 participants were screen failures.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Raltegravir
Number analyzed (Participants) | 37
percent change
  Spine BMD, week 48 (n=37) | 2.7 [1.6 to 3.7]
  Spine BMD, week 96 (n=32) | 3.0 [1.8 to 4.1]
  Total hip BMD week 48 (n=37) | 2.3 [1.4 to 3.1]
  Total hip BMD week 96 (n=32) | 1.9 [1.1 to 2.5]
Statistical Analysis 1: Comparison: Raltegravir; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Percentage of Participants With HIV Viral Load <50 Copies/mL
Description: Plasma HIV viral load remained <50 copies/mL
Time Frame: from Baseline to Week 96
Population: Week 96 data were available for 32 completed participants
Measure: Number; unit: percentage of participants
Arm/Group | Raltegravir
Number analyzed (Participants) | 32
percentage of participants | 90.6

ADVERSE EVENTS:
Time Frame: at 48 and 96 weeks
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Arm/Group | Raltegravir
Serious Adverse Events (participants affected / at risk) | 5/37
Other Adverse Events (participants affected / at risk) | 23/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir (N=37)
PARTNER PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 (1)
RIGHT FLANK/QUADRANT PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
CEREBRAL ANEURYSM (Blood and lymphatic system disorders) | 1 (1)
LEFT KIDNEY STONES (Renal and urinary disorders) | 1 (1)
PROBABLE LUMBAR RADICULOPATHY (Musculoskeletal and connective tissue disorders) | 1 (1)
HOSPITAL ADMISSION FOR MALENA AND FEVERS (Gastrointestinal disorders) | 1 (1)
LOWER REPIRATORY TRACT INFECTION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Raltegravir (N=37)
Abdominal Cramps (Gastrointestinal disorders) | 2
Cold (Respiratory, thoracic and mediastinal disorders) | 2
Conjunctivitis (Eye disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 4
Reflux (Gastrointestinal disorders) | 2
Sleep Apnoea (Respiratory, thoracic and mediastinal disorders) | 2
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 7
Viral Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution, its personnel and the Principal Investigator must not Publish or present any aspect of the Study without the prior written approval of the sponsor. This includes periodic information releases and announcements to the news media or a third party regarding the progress of this Study.